CLINICAL TRIAL: NCT07357129
Title: A Psychosocial Intervention Program to Improve Stress Management Among Young Women: A Pilot Study
Brief Title: Stress Management Intervention for Young Turkish Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bogazici University (Other)
Responsible Party: Principal Investigator, Yasemin Sohtorik İlkmen, Assistant Professor, Bogazici University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-84391427-050.04-258636
Record Dates: First submitted 2026-01-13; First posted 2026-01-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Stress (Psychology)
Keywords: Stress management; pilot study; Self-Help Plus

STUDY DESIGN:
Intervention Model Description: A pilot randomized controlled trial (RCT) will be conducted with a total of 60 participants. Participants will be randomly assigned to one of two groups: 30 individuals will receive the Self-Help Plus (SH+) intervention, while the remaining 30 will not take any intervention and serve as the control group. Upon completion of the intervention sessions and three months after completing the intervention, all participants-including those in the control group-will undergo post-intervention assessments, using the same questionnaires administered at baseline. To ensure ethical considerations and promote equity, the SH+ intervention will be given to control group participants right after the follow-up assessment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Help Plus Intervention Group (Experimental): This arm will receieve Self-Help Plus (SH+) intervention, which is a five-session stress management program developed by the World Health Organization (WHO). The program is designed to be administered in a group format for maximum of 30 participants. Facilitators are not required to be mental health professionals. The best way to implement the program is to train non-specialists from the local communities where it will be delivered. These community members may become facilitators following a brief training. The program is composed of listening to pre-recorded audios along with some group discussions moderated by the facilitators.
  Interventions: Behavioral: Self-Help Plus
- Control Group (No Intervention): Participants in this no intervention group will serve as the control group. Upon the completion of the study (after 3 months follow-up assessments), participants in this group will also receive the same intervention to ensure ethical considerations and promote equity.

INTERVENTIONS:
Behavioral: Self-Help Plus — Self-Help Plus (SH+): SH+ is a five-session stress management program developed by the World Health Organization (WHO). The program is designed to be administered in a group format for maximum of 30 participants. Facilitators are not required to be mental health professionals. The best way to implement the program is to train non-specialists from the local communities where it will be delivered. These community members may become facilitators following a brief training. The program is composed of listening to pre-recorded audios along with some group discussions moderated by the facilitators.
  Arms: Self-Help Plus Intervention Group

SUMMARY:
This pilot study aims to evaluate the feasibility and probable impact of a low intensity psychosocial intervention program designed to help individuals to manage their stress levels. Consequently, this study will implement and measure the feasibility, randomization, retention, assessment procedures, and preliminary effects of the Self-Help Plus (SH+) program developed by the World Health Organization. This intervention, which has been used among immigrants and has proven to be effective, is intended to be implemented for the first time among distressed young Turkish-speaking women in Türkiye (ages between 18 and 29). Participants who will receive this intervention program will be compared with others in the control group who experience similar stress levels but will not receive SH+ during the trial period. Participants in the control group will receive SH+ after the completion of follow-up assessments at 3 months.

DETAILED DESCRIPTION:
This pilot study aims to evaluate the feasibility, acceptability, appropriateness, and probable effectiveness of a community-based stress management program, designed to reduce the stress levels and improve psychological well-being.

Stress is part of daily life; ability to effectively cope with stress plays a crucial role in both physical health and psychological well-being. Numerous studies have shown that effective stress management is a protective factor for physical and psychological well-being. The positive effects of stress coping skills are not limited to reducing current psychological distress; they also act as protective skills, preparing individuals for future stressors. Globally and in Türkiye, the rate of psychiatric disorders is higher among women than men. Major depression and anxiety disorders, the most common disorders around the globe, are twice as common in women as in men.

Consequently, this study aims to implement and measure the feasibility of the Self-Help Plus (SH+) program developed by the World Health Organization in the Turkish context. This intervention, which has been used among immigrants and has proven to be effective, is intended to be implemented for the first time among distressed Turkish-speaking women in Türkiye. The primary goal of the proposed pilot study is to measure its feasibility and probable effectiveness, in order to design a fully powered RCT.

The study will be conducted in Istanbul, Türkiye. Participants will be recruited through social media outlets and via snowballing. Once required number of participants who meet inclusion criteria (distressed without suicide risk) is reached (total of 60 participants), they will be randomly assigned to intervention and control groups (randomization to two arms according to 1:1 principle using an online randomization software). 30 randomly allocated participants will be divided into two groups, and will receive five sessions of SH+ (sessions are weekly, last about 90 to 120 minutes). The remaining 30 participants will be on a waitlist, and will receive the program once follow up assessments are completed. All participants will complete primary and secondary outcome measures at three time points: baseline, within one week upon completion of 5 week sessions (post assessment), and 3 months after the completion of 5 week sessions (follow-up assessment).

ELIGIBILITY:
Inclusion Criteria:

1. being a woman
2. being ages between 18 and 29
3. being fluent in Turkish
4. having high levels of psychological distress (scoring above 15 on the Turkish version of the Kessler Psychological Distress Scale (K-10)

Exclusion Criteria:

1. having an imminent risk of suicide (measured by WHO PM+ assessment tool)
2. having a diagnosis for severe mental disorder (e.g., psychotic disorders or substance dependence)
3. having cognitive impairment (e.g., received a diagnosis of dementia or severe intellectual disability)
4. currently receiving psychological treatment, e.g., therapy.

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants who identify as female
Enrollment: 60 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
K10 | Baseline, within one week after the completion of 5 sessions, and 3 months after the completion of 5 sessions
  Kessler Psychological Distress Scale (K10) is a 10-item questionnaire that aims to measure psychological distress symptoms. Each of the 10 items are scored on a scale of 5 points (1 = "none of the time" to 5= "all of the time"), providing a total score between 10 and 50. Higher scores indicate higher levels of psychological distress. A Turkish version is available and will be used in the current study.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Baseline, within one week of completion of 5 sessions, and 3 months after the completion of 5 sessions
  PHQ-9 is a self-report measure including 9 items that aims to measure the severity of depression symptoms. Each of the 9 items are scored on a 4 point scale (0 = "not at all," to 3= "nearly every day"), providing scores between 0 and 27. Higher scores indicate higher level of depressive symptoms that are related with decreased functional status and increased symptom-related difficulties. Turkish version of the PHQ-9 will be used in the current study.
General Anxiety Disorder-7 (GAD-7) | Baseline, within one week upon completion of 5 sessions, and 3 months after completion of 5 sessions
  GAD-7 is a self-report questionnaire that includes 7 items to measure anxiety symptoms. Each item is scored on a 4 point scale (0 = "not at all," to 3= "nearly every day"), providing scores between 0 and 21. Higher scores indicate higher levels of anxiety. A Turkish version is available, and will be used in the current study.
World Health Organization-Five Well-Being Index (WHO-5) | Baseline, within one week upon completion of 5 sessions, and 3 months after completion of 5 sessions
  Developed by WHO to measure subjective well-being (e.g., calmness and cheerfulness), the WHO-5 consists of a total of 5 questions answered on a 6-point Likert scale (0 = "at no time," to 5 = "all of the time"). Total scores range from zero to 25, higher scores indicating better well-being. The raw total scores are multiplied by four, to generate percentage scores between 0 and 100; percentage scores below 50 are considered to indicate poor mental well-being. The Turkish version will be used in the current study.
General Self Efficacy Scale (GSES) | Baseline, within one week upon completion of 5 sessions, and 3 months after 5 sessions
  GSES is a self-report measure designed to assess the perceived sense of self-efficacy. The scale consists of 10 items rated on a 4-point Likert scale (1 = "not at all true" to 4 = "exactly true"), yielding total scores ranging from 10 to 40. Higher scores indicate higher sense of self-efficacy. The Turkish version will be used in the current study.

IPD SHARING:
Plan to Share IPD: No
Consent for such sharing is not part of the informed consent approved by the ethics committee.

REFERENCES:
- [Background] World Health Organization. "Self-help plus (SH+) training manual". https://iris.who.int/bitstream/handle/10665/379110/9789240095052-eng.pdf?sequence=1 Last Retreived: 8 August 2025.
- [Background] World Health Organization. "Committing to implementation of the Global Strategy for Women's, Children's and Adolescents' Health (2016-2030)". https://iris.who.int/bitstream/handle/10665/366978/WHO-UHL-MCA-GS-23.01-eng.pdf?sequence=1, Last retreived: 8 August 2025.
- [Background] Thoits PA. Stress and health: major findings and policy implications. J Health Soc Behav. 2010;51 Suppl:S41-53. doi: 10.1177/0022146510383499. PMID 20943582
- [Background] Sari, Y. E., Kokoglu, B., Balcioglu, H., Bilge, U., Colak, E. Unluoglu, I. 2016. "Turkish reliability of the patient health questionnaire-9", Biomedical Research-India, 27, S460-S462.
- [Background] Nolen-Hoeksema S. Sex differences in unipolar depression: evidence and theory. Psychol Bull. 1987 Mar;101(2):259-82. No abstract available. PMID 3562707
- [Background] Koyun, A., Taşkın, L., Terzioğlu, F. 2011. "Yaşam dönemlerine göre kadın sağlığı ve ruhsal işlevler: Hemşirelik yaklaşımlarının değerlendirilmesi", Psikiyatride Güncel Yaklaşımlar, 3(1), 67-99.
- [Background] Min JA, Lee CU, Lee C. Mental health promotion and illness prevention: a challenge for psychiatrists. Psychiatry Investig. 2013 Dec;10(4):307-16. doi: 10.4306/pi.2013.10.4.307. Epub 2013 Dec 16. PMID 24474978
- [Background] Konkan, R., Senormanci, O., Guclu, O., Aydin, E. Sungur, M. Z., 2013. "Validity and reliability study for the Turkish adaptation of the Generalized Anxiety Disorder-7 (GAD-7) scale/Yaygin Anksiyete Bozuklugu-7 (YAB-7) testi Turkce uyarlamasi, gecerlik ve güvenirliği", Archives of Neuropsychiatry, 50(1), 53-59.
- [Background] Kessler RC, Barker PR, Colpe LJ, Epstein JF, Gfroerer JC, Hiripi E, Howes MJ, Normand SL, Manderscheid RW, Walters EE, Zaslavsky AM. Screening for serious mental illness in the general population. Arch Gen Psychiatry. 2003 Feb;60(2):184-9. doi: 10.1001/archpsyc.60.2.184. PMID 12578436
- [Background] Eser E, Cevik C, Baydur H, Gunes S, Esgin TA, Oztekin CS, Eker E, Gumussoy U, Eser GB, Ozyurt B. Reliability and validity of the Turkish version of the WHO-5, in adults and older adults for its use in primary care settings. Prim Health Care Res Dev. 2019 Jul 1;20:e100. doi: 10.1017/S1463423619000343. PMID 32800004
- [Background] Dil, S. 2017. "Kadın ruh sağlığı epidemiyolojik göstergeleri ve toplumsal cinsiyet", Turkiye Klinikleri J Psychiatr Nurs-Special Topics, 3(3), 198-203.
- [Background] Aypay, A. 2010. "The Adaptation Study of General Self-Efficacy (GSE) Scale to Turkish", Inonu University Journal of the Faculty of Education (INUJFE), 11(2).
- [Background] Acarturk C, Uygun E, Ilkkursun Z, Carswell K, Tedeschi F, Batu M, Eskici S, Kurt G, Anttila M, Au T, Baumgartner J, Churchill R, Cuijpers P, Becker T, Koesters M, Lantta T, Nose M, Ostuzzi G, Popa M, Purgato M, Sijbrandij M, Turrini G, Valimaki M, Walker L, Wancata J, Zanini E, White RG, van Ommeren M, Barbui C. Effectiveness of a WHO self-help psychological intervention for preventing mental disorders among Syrian refugees in Turkey: a randomized controlled trial. World Psychiatry. 2022 Feb;21(1):88-95. doi: 10.1002/wps.20939. PMID 35015365
- See also: WHO: Committing to implementation of the Global Strategy for Women's, Children's and Adolescents' Health (2016-2030) — https://iris.who.int/bitstream/handle/10665/366978/WHO-UHL-MCA-GS-23.01-eng.pdf?sequence=1